CLINICAL TRIAL: NCT00198822
Title: Impact of Maternal Vitamin A or Beta-Carotene Supplementation on Maternal and Infant Mortality in Bangladesh
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: United States Agency for International Development (USAID) (U.S. Federal Agency); Bill and Melinda Gates Foundation (Other); Canadian International Development Agency (Other Government); The Sight and Life Research Institute (Unknown); Access Business Group (Industry)
Responsible Party: Principal Investigator, Keith P. West, Professor, Johns Hopkins Bloomberg School of Public Health
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: GHS-A-00-03-00019-00
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Results first posted 2011-10-12 (Estimated); Last update posted 2012-03-07 (Estimated); Status verified 2012-03

CONDITIONS: Vitamin A Deficiency; Maternal Mortality; Infant Mortality
Keywords: Maternal mortality; Infant mortality; Vitamin A; Beta-carotene; Micronutrients; Bangladesh; Neonatal mortality
MeSH Terms: conditions — Vitamin A Deficiency; Maternal Death; Infant Death | interventions — Vitamin A

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): Weekly oral supplement with 7000 µg retinol equivalents from early pregnancy through 12 weeks following termination of pregnancy
  Interventions: Dietary Supplement: Vitamin A or Beta-Carotene Supplements
- 2 (Experimental): Weekly oral supplement with 42 mg of beta-carotene from early pregnancy through 12 weeks following termination of pregnancy
  Interventions: Dietary Supplement: Vitamin A or Beta-Carotene Supplements
- 3 (Placebo Comparator): Weekly oral supplement with placebo from early pregnancy through 12 weeks following termination of pregnancy
  Interventions: Dietary Supplement: Vitamin A or Beta-Carotene Supplements

INTERVENTIONS:
Dietary Supplement: Vitamin A or Beta-Carotene Supplements — weekly dosage of either 7000 µg retinol equivalents as preformed vitamin A or 42 mg of beta-carotene from 1st trimester of pregnancy through 12 weeks after termination of pregnancy

SUMMARY:
The purpose of this trial is to determine whether providing women with a weekly oral supplement of vitamin A, either preformed or as beta-carotene, at a dosage equivalent to a recommended intake from early pregnancy through three months postpartum, can reduce the risk of maternal mortality, fetal loss, or infant mortality.

DETAILED DESCRIPTION:
Maternal mortality and vitamin A deficiency coexist in rural South Asia. In Nepal, weekly supplementation with vitamin A or beta-carotene during the child-bearing years reduced all-cause maternal mortality and, in night blind women, also infant mortality. The present trial is testing the efficacy of the same supplements from ~9 weeks' gestation to 12 weeks postpartum. The planned sample size is 68,000 pregnancies. It is being conducted in 19 rural unions, covering an area of ~750 sq km with a population of ~580,000 in Gaibandha and Southern Rangpur Districts in Northern Bangladesh. The study area was mapped as 596 "sectors" (unit of randomization), each comprising 200-275 households; ~135,000 houses were numerically addressed and, at the outset, 103,000 women were listed. Women are visited at home every 5 weeks by 596 trained female staff to detect pregnancy by a combination of menstrual history and urine testing. Newly married women are prospectively enlisted for pregnancy surveillance. Following informed consent urine-positive (pregnant) women detected during surveillance are enrolled to receive weekly a capsule containing 7000 retinol equivalents of preformed vitamin A, 42 mg of beta-carotene or placebo. Vital events are recorded weekly through 3 months postpartum. Trained interviewers conduct maternal nutritional and health and household socioeconomic assessments in the 1st trimester. At 3 months postpartum, interviewers assess both mother and infant for health and nutritional status, including apparent birth defects that are later physician-confirmed. An additional home health assessment occurs at 6 months post partum, and vital status is recorded for mother and infant at one year postpartum. A ~3% subsample of enrolled pregnant women participate in a substudy involving enhanced clinical, anthropometric, biochemical, body compositional, morbidity and interview-based assessment protocols in the 1st, 2nd and 3rd trimesters, and at 3 months post-partum. Reported maternal and infant deaths are verified and causes ascertained during "verbal autopsy" interviews with family members of the deceased.

ELIGIBILITY:
Inclusion Criteria:

* Married women of reproductive age
* First pregnancy during time period of trial

Exclusion Criteria:

* Premenarchial girls
* Married women with a previous pregnancy enrolled into the trial
* Previously married women who have moved into the study area
* Single women (never married, widowers)
* Women who are sterilized (or whose husbands are sterilized)
* Menopausal women

Ages: 15 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 59666 (Actual)
Dates: Start 2001-08; Primary Completion 2007-01 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Keith P West, Jr., Dr.P.H., Principal Investigator — Johns Hopkins Bloomberg School of Public Health; Parul Christian, Dr.P.H., Study Director — Johns Hopkins Bloomberg School of Public Health; Rolf DW Klemm, Dr.P.H., Study Director — Johns Hopkins Bloomberg School of Public Health; Mahbubur Rashid, MBBS, MSc, Study Director — JiVitA Bangladesh Project; Alain B Labrique, MSc, Study Director — Johns Hopkins Bloomberg School of Public Health; Alfred Sommer, M.D., Study Director — Johns Hopkins Bloomberg School of Public Health
Locations (3):
- Johns Hopkins School of Public Health, Baltimore, Maryland, United States
- Bangladesh (2):
  - JiVitA Bangladesh Project, Rangpur, Rajshahi Division
  - JiVitA Project Office, Rangpur City, Rangpur District

REFERENCES:
- [Background] West KP Jr, Katz J, Khatry SK, LeClerq SC, Pradhan EK, Shrestha SR, Connor PB, Dali SM, Christian P, Pokhrel RP, Sommer A. Double blind, cluster randomised trial of low dose supplementation with vitamin A or beta carotene on mortality related to pregnancy in Nepal. The NNIPS-2 Study Group. BMJ. 1999 Feb 27;318(7183):570-5. doi: 10.1136/bmj.318.7183.570. PMID 10037634
- [Background] Katz J, West KP Jr, Khatry SK, Pradhan EK, LeClerq SC, Christian P, Wu LS, Adhikari RK, Shrestha SR, Sommer A. Maternal low-dose vitamin A or beta-carotene supplementation has no effect on fetal loss and early infant mortality: a randomized cluster trial in Nepal. Am J Clin Nutr. 2000 Jun;71(6):1570-6. doi: 10.1093/ajcn/71.6.1570. PMID 10837300
- [Background] Christian P, West KP Jr, Khatry SK, LeClerq SC, Kimbrough-Pradhan E, Katz J, Shrestha SR. Maternal night blindness increases risk of mortality in the first 6 months of life among infants in Nepal. J Nutr. 2001 May;131(5):1510-2. doi: 10.1093/jn/131.5.1510. PMID 11340108
- [Background] Christian P, West KP Jr, Khatry SK, Katz J, LeClerq SC, Kimbrough-Pradhan E, Dali SM, Shrestha SR. Vitamin A or beta-carotene supplementation reduces symptoms of illness in pregnant and lactating Nepali women. J Nutr. 2000 Nov;130(11):2675-82. doi: 10.1093/jn/130.11.2675. PMID 11053506
- [Background] Christian P, West KP Jr, Khatry SK, Kimbrough-Pradhan E, LeClerq SC, Katz J, Shrestha SR, Dali SM, Sommer A. Night blindness during pregnancy and subsequent mortality among women in Nepal: effects of vitamin A and beta-carotene supplementation. Am J Epidemiol. 2000 Sep 15;152(6):542-7. doi: 10.1093/aje/152.6.542. PMID 10997544
- [Background] West KP Jr. Extent of vitamin A deficiency among preschool children and women of reproductive age. J Nutr. 2002 Sep;132(9 Suppl):2857S-2866S. doi: 10.1093/jn/132.9.2857S. PMID 12221262
- [Result] West KP Jr, Christian P, Labrique AB, Rashid M, Shamim AA, Klemm RD, Massie AB, Mehra S, Schulze KJ, Ali H, Ullah B, Wu LS, Katz J, Banu H, Akhter HH, Sommer A. Effects of vitamin A or beta carotene supplementation on pregnancy-related mortality and infant mortality in rural Bangladesh: a cluster randomized trial. JAMA. 2011 May 18;305(19):1986-95. doi: 10.1001/jama.2011.656. PMID 21586714
- [Result] Labrique AB, Christian P, Klemm RD, Rashid M, Shamim AA, Massie A, Schulze K, Hackman A, West KP Jr. A cluster-randomized, placebo-controlled, maternal vitamin A or beta-carotene supplementation trial in Bangladesh: design and methods. Trials. 2011 Apr 21;12:102. doi: 10.1186/1745-6215-12-102. PMID 21510905
- [Result] Gunnsteinsson S, Labrique AB, West KP Jr, Christian P, Mehra S, Shamim AA, Rashid M, Katz J, Klemm RD. Constructing indices of rural living standards in Northwestern Bangladesh. J Health Popul Nutr. 2010 Oct;28(5):509-19. doi: 10.3329/jhpn.v28i5.6160. PMID 20941903
- [Derived] Surkan PJ, Sakyi KS, Christian P, Mehra S, Labrique A, Ali H, Ullah B, Wu L, Klemm R, Rashid M, West KP Jr, Strobino DM. Risk of Depressive Symptoms Associated with Morbidity in Postpartum Women in Rural Bangladesh. Matern Child Health J. 2017 Oct;21(10):1890-1900. doi: 10.1007/s10995-017-2299-7. PMID 28766094
- [Derived] Ali H, Hamadani J, Mehra S, Tofail F, Hasan MI, Shaikh S, Shamim AA, Wu LS, West KP Jr, Christian P. Effect of maternal antenatal and newborn supplementation with vitamin A on cognitive development of school-aged children in rural Bangladesh: a follow-up of a placebo-controlled, randomized trial. Am J Clin Nutr. 2017 Jul;106(1):77-87. doi: 10.3945/ajcn.116.134478. Epub 2017 May 10. PMID 28490513
- [Derived] Sundaram ME, Ali H, Mehra S, Shamim AA, Ullah B, Rashid M, Shaikh S, Christian P, Klemm RD, West KP Jr, Labrique A. Early newborn ritual foods correlate with delayed breastfeeding initiation in rural Bangladesh. Int Breastfeed J. 2016 Dec 8;11:31. doi: 10.1186/s13006-016-0090-9. eCollection 2016. PMID 27980605
- [Derived] Surkan PJ, Sakyi K, Strobino DM, Mehra S, Labrique A, Ali H, Ullah B, Wu L, Klemm R, Rashid M, West KP, Christian P. Depressive symptoms in mothers after perinatal and early infant loss in rural Bangladesh: a population-based study. Ann Epidemiol. 2016 Jul;26(7):467-473. doi: 10.1016/j.annepidem.2016.06.001. Epub 2016 Jun 8. PMID 27449568
- [Derived] Shamim AA, Schulze K, Merrill RD, Kabir A, Christian P, Shaikh S, Wu L, Ali H, Labrique AB, Mehra S, Klemm RD, Rashid M, Sungpuag P, Udomkesmalee E, West KP Jr. First-trimester plasma tocopherols are associated with risk of miscarriage in rural Bangladesh. Am J Clin Nutr. 2015 Feb;101(2):294-301. doi: 10.3945/ajcn.114.094920. Epub 2014 Nov 26. PMID 25646326
- [Derived] Christian P, Klemm R, Shamim AA, Ali H, Rashid M, Shaikh S, Wu L, Mehra S, Labrique A, Katz J, West KP Jr. Effects of vitamin A and beta-carotene supplementation on birth size and length of gestation in rural Bangladesh: a cluster-randomized trial. Am J Clin Nutr. 2013 Jan;97(1):188-94. doi: 10.3945/ajcn.112.042275. Epub 2012 Nov 14. PMID 23151532
- [Derived] Christian P, Labrique AB, Ali H, Richman MJ, Wu L, Rashid M, West KP Jr. Maternal vitamin A and beta-carotene supplementation and risk of bacterial vaginosis: a randomized controlled trial in rural Bangladesh. Am J Clin Nutr. 2011 Dec;94(6):1643-9. doi: 10.3945/ajcn.111.019059. Epub 2011 Nov 9. PMID 22071710
- [Derived] Shamim AA, Christian P, Schulze KJ, Ali H, Kabir A, Rashid M, Labrique A, Salamatullah Q, West KP Jr. Iodine status in pregnancy and household salt iodine content in rural Bangladesh. Matern Child Nutr. 2012 Apr;8(2):162-73. doi: 10.1111/j.1740-8709.2010.00282.x. Epub 2010 Oct 26. PMID 20977661

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Women were recruited into the trial from August 2001 to January 2007. As this was a community trial, we identified pregnant women by conducting a urine test on women reporting to be amenstrual from the last visit during 5 weekly visit cycles to their homes in rural communities of the districts of Rangpur and Gaibandha, Bangladesh.
Groups:
- 1 Placebo Control: Weekly oral supplement with placebo from early pregnancy through 12 weeks following termination of pregnancy
- 2 Vitamin A Supplement: Weekly oral supplement with 7000 micrograms of retinol equivalents from early pregnancy through 12 weeks following termination of pregnancy
- 3 Beta-Carotene Group: Weekly oral supplement with 42 mg of all-trans beta-carotene from early pregnancy through 12 weeks following termination of pregnancy
Period: Overall Study
Arm/Group | 1 Placebo Control | 2 Vitamin A Supplement | 3 Beta-Carotene Group
Started | 19876 (No. of consenting pregnant women in the placebo arm of trial cohort) | 19826 (No. of consenting pregnant women in the vitamin A arm of trial cohort) | 20019 (No. of consenting pregnant women in the beta-catorene arm of trial cohort)
Completed | 19862 (No. of consented pregnant women in placebo arm with vital status known at 12 weeks postpartum) | 19806 (No. of consented pregnant women in vitamin A arm with vital status known at 12 weeks postpartum) | 19998 (No. of consented pregnant women in beta-catorene arm with vital status known at 12 weeks postpartum)
Not Completed | 14 | 20 | 21
Not completed — Lost to Follow-up | 14 | 20 | 21

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1 Placebo Control | 2 Vitamin A Supplement | 3 Beta-Carotene Group | Total
Number analyzed (Participants) | 19862 | 19806 | 19998 | 59666
Age Categorical [Number; unit: participants] — A very small number of women in the study were unable to recollect or even work out their age. In rural South Asia, this is not uncommon and of the 35 women for whom we do not have an age, 14 are in the placebo group, 15 in the Vitamin A group and 6 in the beta-carotene group.
  participants
    <=18 years | 5875 | 5774 | 5936 | 17585
    Between 18 and 65 years | 13973 | 14017 | 14056 | 42046
    >=65 years | 0 | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] — A very small number of women in the study were unable to recollect or even work out their age. In rural South Asia, this is not uncommon and of the 35 women for whom we do not have an age, 14 are in the placebo group, 15 in the Vitamin A group and 6 in the beta-carotene group.
  years | 23.03 (6.53) | 23.17 (6.56) | 23.06 (6.56) | 23.09 (6.55)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19862 | 19806 | 19998 | 59666
  Male | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Bangladesh | 19862 | 19806 | 19998 | 59666

OUTCOME MEASURES:

1. Secondary Outcome: All-cause 3-month Infant Mortality
Time Frame: Deaths through the 1st 12 weeks of life
Population: Mortality evaluated on intent-to-treat basis
Measure: Number; unit: participants
Arm/Group | 1 Placebo Control | 2 Vitamin A Supplement | 3 Beta-Carotene Group
Number analyzed (Participants) | 13965 | 13898 | 14018
participants | 951 | 904 | 979

2. Secondary Outcome: Maternal Morbidity, Including Obstetric Complications
Time Frame: through the 1st 24 weeks following termination of pregnancy
Reporting Status: Not Posted

3. Secondary Outcome: Gestational Age at Birth
Time Frame: within 24 weeks after birth
Reporting Status: Not Posted

4. Secondary Outcome: Fetal Growth and Postnatal Infant Growth Through Three Months of Age
Time Frame: through the 1st 12 weeks after birth
Reporting Status: Not Posted

5. Secondary Outcome: Infant Morbidity Through 3 Months of Age
Time Frame: within 24 weeks after birth
Reporting Status: Not Posted

6. Secondary Outcome: Plasma Beta-carotene in the Third Trimester of Pregnancy(Nutritonal Status of the Mother)
Time Frame: Third trimester of pregnancy (about the 32nd week of gesatation)
Measure: Mean (Standard Deviation); unit: Plasma beta-carotene micromoles / liter
Arm/Group | 1 Placebo Control | 2 Vitamin A Supplement | 3 Beta-Carotene Group
Number analyzed (Participants) | 332 | 367 | 368
Plasma beta-carotene micromoles / liter | 0.11 (0.09) | 0.12 (0.12) | 0.12 (0.10)

7. Primary Outcome: All-cause, Pregnancy-related Mortality
Description: Mortality evaluated on intent-to-treat basis
Time Frame: Deaths during pregnancy through 12 weeks postpartum
Population: As the study ended on the advice of the Data and Safety Monitoring Board, based on evidence of no difference, all enrolled women who had a chance of being followed through 84 days after the end of their pregnancy were included in the trial. The cohort included pregnancies identified between August 17, 2001 and January 5, 2006.
Measure: Number; unit: Participants
Arm/Group | 1 Placebo Control | 2 Vitamin A Supplement | 3 Beta-Carotene Group
Number analyzed (Participants) | 19862 | 19806 | 19998
Participants | 41 | 47 | 50
Statistical Analysis 1: Comparison: 1 Placebo Control vs 2 Vitamin A Supplement vs 3 Beta-Carotene Group; Sample size was based on an expected placebo group MR of 600/100,000 pregnancies, requiring 18,000 pregnancies to detect a 35% reduction in all-cause mortality, with a 5% type I error, 80% power, 1.21 design effect, 15% early pregnancy loss and 10% loss to follow-up. A mid-study DSMB analysis suggested a lower MR, leading the SS to be increased to 67,740. However, with no mortality difference evident at a DSMB meeting in Dec 2006, the trial was halted leaving 59,721 in the trial cohort; Test type: Superiority or Other; p = 0.05, generalized estimating equations — We set an a priori level of statistical significance of p equal to 0.05; RR with 95% CIs were estimated by GEE binomial regression, with a log link function and exchangeable correlation appropriate for binary data; Risk Ratio (RR) = 0.65, 95% CI 1-sided [upper limit 0.99] — The vitamin A group and the Beta-carotene group were compared to the placebo group

8. Secondary Outcome: Plasma Retinol at the Third Trimester of Pregnancy (Nutritional Status of the Mother)
Time Frame: Third trimester of pregnancy (about the 32nd week of gestation)
Measure: Mean (Standard Deviation); unit: micromoles per liter
Arm/Group | 1 Placebo Control | 2 Vitamin A Supplement | 3 Beta-Carotene Group
Number analyzed (Participants) | 332 | 367 | 368
micromoles per liter | 1.02 (0.31) | 1.25 (0.33) | 1.06 (0.33)

ADVERSE EVENTS:
Arm/Group | 1 Placebo Control | 2 Vitamin A Supplement | 3 Beta-Carotene Group
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No